CLINICAL TRIAL: NCT00390546
Title: Multicenter Study of Antiarrhythmic Medications for Treatment of Infants With Supraventricular Tachycardia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Hospital for Sick Children (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Shubhayan Sanatani, principal investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H06-70156
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Digoxin; Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Propranolol (Experimental): Single dose of 0.5 mg/kg per dose and increased to 1.0 mg/kg per dose ITD for the second and subsequent doses.
  Interventions: Drug: Propranolol
- Digoxin (Experimental): First 2 doses at 0.010 mg/kg per dose TID, then 0.0035 mg/kg per dose TID for the third and subsequent doses
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin
  Arms: Digoxin
Drug: Propranolol
  Arms: Propranolol

SUMMARY:
This is a randomized, double-blind, multi-centered study to compare 6 months of medical treatment with digoxin or propranolol in infants with SVT Background: SVT is the most common sustained arrhythmia of infancy. Neither digoxin nor propranolol has been evaluated for pediatric use in a controlled trial in the context of SVT, yet both medications are used frequently.

Specific aims of the study:

To determine whether propranolol and digoxin differ in the:

1. Incidence of recurrent SVT in infants after 6 months of treatment with propranolol or digoxin
2. Time to first recurrence of SVT in infants treated with propranolol or digoxin.
3. Incidence of adverse outcomes in infants treated with propranolol or digoxin.

DETAILED DESCRIPTION:
The purpose of the proposed research is to conduct a randomized double-blind, multi-centre study of two antiarrhythmic medications, digoxin and propranolol, to evaluate whether one of these medications is more effective in reducing risk of recurrent supraventricular tachycardia (SVT) in infants.

SVT is the most common sustained arrhythmia of infancy, occurring in 1 in 250-1000 children, and is a serious health burden in Canada and internationally [1, 5-8]. SVT is a common clinical problem facing many health care providers, including general pediatricians, emergency room physicians, nurses, cardiologists, and intensive care physicians. SVT carries significant morbidity and mortality, and patients typically receive long-term medical therapy. Untreated, an infant can tolerate SVT for only a short period before heart failure and shock (or even death) ensues. The management of SVT is currently under debate and often appears to depend on physician preference [9]. While spontaneous termination of the acute episode may occur [1, 2, 6, 9, 10], many infants require medical intervention to terminate the episode. Vagal maneuvres and adenosine have reasonable success in terminating an acute SVT episode, but other medications may also be required. Once the acute episode is treated, the physician(s) must make a decision whether or not to start maintenance (chronic) therapy.

At present, there is no clinical consensus for the management of SVT in infancy. The rationale for chronic therapy in SVT is to prevent recurrences and to limit symptoms during recurrences. Yet SVT recurrences are not readily predictable [11]. Many medications are available to treat SVT; however, these medications have associated risks and there are psychosocial implications for families. To date, most medications used to treat infant SVT have not been evaluated in controlled studies of infants. Thus, at present, physicians must make decisions about initiation and duration of chronic therapy and choice of medication in the absence of evidence from controlled clinical trials. A prospective, randomized clinical study is crucial to provide evidence to guide therapy of infant SVT.

As a preliminary study to inform the proposed trial, we carried out a survey of all pediatric cardiologists in North America [12]. In this survey, we presented hypothetical cases of infants with SVT and asked about acute and chronic management. Several points are clear:

* 11 different medications were chosen for the management of infant SVT;
* there was a discrepancy among respondents with respect to medication choices, based on whether the respondent had additional electrophysiology training or not; and
* several physicians selected digoxin in infants who have Wolff-Parkinson-White syndrome ; this medication choice may have deleterious effects in these infants.

Our survey identified that, among the wide range of medications used to manage infant SVT, the two most commonly used ones are digoxin and propranolol. Digoxin and propranolol are both well established, widely used medications in both infants and adults. Eighty-five percent of survey respondents reported using one or both to manage infant SVT, but did not rationalize their choice nor determine whether one or the other is better to reduce risk of SVT recurrence or whether one is associated with fewer adverse events. Furthermore, pediatric cardiologists and electrophysiologists differed in medication choice.

Thus, to provide evidence to improve clinical decision-making and infant health, we propose to conduct a prospective, randomized double-blind, multi-centre study of digoxin and propranolol for treatment of infant SVT.

The specific aims of the proposed trial are to determine whether these medications differ in the:

1. Incidence of recurrent SVT in infants after 6 months of treatment with propranolol or digoxin;
2. Time to first recurrence of SVT in infants treated with propranolol or digoxin;
3. Incidence of adverse outcomes in infants treated with propranolol or digoxin. BACKGROUND SUPRAVENTRICULAR TACHYCARDIA In infants and children, SVT results primarily from an accessory connection between the atrium and ventricle [5, 8-10, 13]. This provides the substrate for a reentrant circuit utilizing the normal conduction system and the accessory pathway, resulting in an atrioventricular reciprocating tachycardia (AVRT). A similar reentrant circuit can exist within the atrioventricular node, resulting in an atrioventricular nodal reentrant tachycardia (AVNRT); however, this is much less common in infants [5, 13, 14]. Both AVRT and AVNRT result in a very rapid heart rate with an attendant decrease in diastolic filling time and cardiac output. The differentiation of these two mechanisms is not always easily made on the surface electrocardiogram (ECG) [8, 15], and currently the same therapies are applied for both conditions [16].

Most cases (61-73%) of infant SVT occur by age 4 months [9, 17, 18], and almost all occur before the age of 12 months [1, 2, 5, 6, 9, 13, 17-19]. In 1981, Garson et al. reported data from one of the largest retrospective series, encompassing 217 SVT referrals over 25 years [6]. Infants who presented with SVT before 4 months of age had faster tachycardia rates and a greater risk of presenting with congestive heart failure (CHF) (24%) than did older infants or children. Although infants can tolerate SVT for >24 hours before signs of CHF ensue [1], CHF is seen in a significant number of patients (24-54%) when they come to medical attention. Infants with CHF can progress to cardiovascular collapse, accounting for the mortality of 1-4% in infants with SVT [2, 5, 6, 20].

The acute management of infant SVT is debated and often depends on physician preference [9]. In 9-50% of cases, the acute SVT episode ends spontaneously [1, 2, 6, 9, 10] and in 70-90% of patients, adenosine and/or vagal maneuvres (e.g. applying ice pack to the face) work with reasonable success; however, other medications (e.g. amiodarone) may also be required [1, 2, 8, 9]. Once the acute episode is over, the physician and family must make a decision about whether or not to start chronic therapy.

SVT RECURRENCE & CHRONIC THERAPY The rationale for chronic therapy in SVT is to prevent recurrences and to limit symptoms during recurrences [8]. SVT can be repetitive, but the recurrences are not readily predictable [11]. There is a wide range-from 0% to 78%-of reported recurrences of SVT, even with medical treatment [1, 2, 6, 19, 21]. There are several studies with reliable data (see Table 1 at end), but some reports of the predictors of recurrent episodes may include data that are not applicable to all patients and may involve invasive studies [21-23]. The physician attitude towards chronic therapy has also changed. While in Garson's 1981 study, chronic medication was started in only 72% of cases, our survey indicated that 98% of respondents would initiate chronic therapy [12]. This likely reflects the goal of minimizing morbidity and mortality in the care of all children with heart disease. In Garson's review, recurrences were common (56%) and most (75%) occurred within 3 months of the initial SVT presentation [6]. Perry et al. observed that, in 60 patients who presented by 2 months of age, SVT had disappeared in 93% by 8 months of age, but many had recurrences later in life [19]. Tortoriello found that patients without pre-excitation had a low (17%) risk of recurrence [4].

Our knowledge of the natural history of infants with SVT is incomplete, both in terms of the need for chronic therapy and the duration. Despite the fact that the risk of recurrence is not known (and may be <50%), due to the potential for serious adverse outcomes, most pediatric cardiologists advocate chronic therapy after an infant presents with SVT. The early clinical course can be variable, but most patients do not require medical therapy beyond the first few months of life [7, 20]. The duration of therapy has ranged over the studies but currently lasts 6 to 12 months after presentation [6, 9] because of the uncertainties of the clinical course [20, 24, 25]. The risk of recurrence during the first year of life has not been determined definitively.

THE MEDICATIONS Chronic therapy for SVT usually entails daily antiarrhythmic medication (see Table 2 below). Currently, choice of medication is guided by retrospective reviews, rather than by controlled trials [3-6, 16, 17, 26]. Our survey identified that, among the wide range of medications used to manage infant SVT, the most commonly used are digoxin and propranolol [12].

Table 2. Commonly used medications for the chronic treatment of supraventricular tachycardia Digoxin Propranolol Sotalol Amiodarone Flecainide Propafenone Verapamil Atenolol Nadolol Digoxin is a sodium-potassium exchange pump inhibitor that has neuro-humoral effects and effects on cardiac conduction. Its efficacy as an antiarrhythmic drug is attributed to direct atrioventricular nodal blocking properties, combined with parasympathetic (vagal) activation, which slows sinus rate, decreases conduction velocity, and increases atrioventricular nodal refractoriness. For decades, digoxin has been reported to be the preferred medication to prevent recurrence of SVT in infants [1, 2], and it remains a common choice [3, 4]. In one retrospective review of 26 cases of infant SVT, Pfammatter & Stockler found that 65% had no recurrences on prophylactic digoxin therapy [3]. Deal et al reported that 61% of infants were treated with digoxin and that 37% of this group required additional or combination therapy, most commonly with propranolol [2].

Propranolol is a non-selective beta-adrenergic blocker that has some sodium blockade, but primarily exerts its antiarrhythmic effects through antagonism of catecholamine-mediated effects on cardiac conduction. This antagonism results in slowed conduction velocity, increased refractoriness, and reduced automaticity, especially in sinoatrial and atrioventricular nodal tissue. Propranolol is also reported to be effective in SVT [17]. Retrospective reviews have not always found differences in recurrence rates among infants treated with digoxin versus propranolol: some report equal efficacy in preventing recurrent SVT [4, 5, 17], while others report a lower recurrence with propranolol [27-29].

Digoxin and propranolol have a wide range of reported efficacy for preventing recurrence of SVT [5, 17] and neither digoxin nor propranolol is fully effective; treatment failures can reach 26% [17] and additional antiarrhythmics are often required [4, 8, 16, 26, 30-36]. Digoxin and propranolol are often referred to as "first-line agents", i.e. the medications that will be started initially to prevent recurrences of SVT. Several studies have reported on the use of medications in combination without specifying details (see Table 1). There are limited data on side effect profiles of digoxin and propranolol [16, 37, 38]. Despite this lack of data, digoxin and propranolol are used over other agents whose side effect profiles have been the subject of greater scrutiny, perhaps due to their relative "newness" [30-33, 35, 36, 39]. Both are frequently used for chronic therapy of infant SVT, but they have never been compared in a controlled trial.

WHY THE TRIAL IS NEEDED NOW Management of infant SVT is confounded by several factors, including the variable clinical course, the inability to predict recurrence, and the 'unknown' natural history in terms of resolution of arrhythmia substrate. This creates a challenge for health care practitioners and families. Our preliminary survey demonstrated a discrepancy between pediatric electrophysiologists and pediatric cardiologists in their medication choice for treatment of infant SVT [12]. It is not clear why the 'experts' (the electrophysiologists) manage SVT differently than do the majority of physicians who see infants with SVT. Most importantly, these treatment decisions are being made without clear evidence to support these choices. The differences in medication choice may reflect concern over case reports of rapid conduction and atrial arrhythmias with digoxin use in the setting of Wolff-Parkinson-White syndrome [2, 9, 27, 40]. It may be that electrophysiologists do not choose digoxin because of reports of high recurrence rates [10, 20, 26]; it is not clear whether digoxin poses a risk in the first year of life [17, 41]. Propranolol is reported to be effective at preventing recurrences and continues to be recommended for use [2, 6, 16]. Furthermore, interpretation of the existing body of knowledge poses several limitations. For example, almost all studies of SVT in childhood are retrospective in nature, spanning many years, and include studies of patients with varying forms of SVT, including those with Wolff-Parkinson-White syndrome and those with structural heart disease. In many cases, treatment failures and successes are not defined consistently, and multiple medication regimens are common. At the conclusion of these studies, reference is frequently made to the need for a controlled clinical trial. The lack of controlled trial outcomes, in turn, is cited as a key limitation for interpreting existing published data [8, 26].

The Health Protection Branch of Health Canada and The Food and Drug Administration of the United States both recognize the need for controlled clinical trials in pediatric patients. To our knowledge, neither digoxin nor propranolol has been evaluated for pediatric use in a controlled trial in the context of SVT, yet both medications are used frequently. Therefore, this study is needed because digoxin and propranolol continue to be used as the most common therapy for prevention of recurrent SVT. There is a significant debate about their effectiveness, with a division between experts in the field and general cardiologists. There may be a large impact on patients if one medication is better than the other or has more adverse outcomes (e.g. hospital admissions). The results of this trial have significant potential for direct impact on infant health and provision of care in Canada and globally. This is evidenced by the large number of electrophysiologists endorsing the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Presentation with SVT due to AVRT or AVNRT.
2. Age 4 months or less at presentation.
3. No major structural heart disease (patent foramen ovale and patent ductus arteriosus are allowable.
4. No other significant co-morbid condition likely to result in non-compliance or death in next 6 months.

The SVT mechanism will be presumed to be AVRT or AVNRT if the ECG shows:

* Normal complex tachycardia with abrupt onset and offset;
* The RR interval remains relatively constant during tachycardia with heart rates of 220-310 bpm;
* VA (ventriculo-atrial) association [i.e., there is a 1:1 AV relationship (except for cases of proven AV nodal reentry with a 2:1 relationship between atrium and ventricle)]; and
* Termination of tachycardia with vagal maneuvres or adenosine with AV block or VA block.

Additional supportive information:

* The presence of a P wave in either the ST segment or T wave, or the presence of a P wave altering the terminal portion of the QRS complex;
* Spontaneous termination of the tachycardia with a P wave;
* Onset with prolongation of the PR interval;
* Altered rate with resolution of temporary bundle branch block;
* Esophageal or electrophysiology study confirming tachycardia mechanism.

Exclusion Criteria:

1. Failure to obtain consent;
2. Known hypersensitivity to either study medication or suspension;
3. Structural heart disease other than a patent foramen ovale or patent ductus arteriosus;
4. Persistent abnormal cardiac function documented by echocardiogram (shortening fraction <28%) in sinus rhythm;
5. Pre-excitation (Wolff Parkinson White syndrome);
6. Permanent junctional reciprocating tachycardia;
7. Ectopic atrial tachycardia;
8. Atrial flutter;
9. Sick sinus syndrome or significant bradycardia;
10. Long QT syndrome;
11. Digoxin > 40 micrograms/kg total received within past 7 days
12. Amiodarone >50 milligrams/kg total received within past month
13. Asthma or obstructive airway disease;
14. Renal failure.

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2006-10; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shubhayan Sanatani, MD, Principal Investigator — University of British Columbia
Locations (14):
- United States (10):
  - University of Southern California - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Schneider Children's Hospital, New Hyde Park, New York
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital Ohio, Columbus, Ohio
  - Medical University of Charleston South Carolina, Charleston, South Carolina
  - Primary Children's Medical Centre, Salt Lake City, Utah
  - Norfolk Children's Hospital of the King's Daughter's, Norfolk, Virginia
  - Northwest Pediatric Cardiology, Spokane, Washington
- Canada (4):
  - Stollery children's Hospital, Edmonton, Alberta
  - Sonia Franciosi, Vancouver, British Columbia
  - Hospital for Sick Kids, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Sanatani S, Potts JE, Reed JH, Saul JP, Stephenson EA, Gibbs KA, Anderson CC, Mackie AS, Ro PS, Tisma-Dupanovic S, Kanter RJ, Batra AS, Fournier A, Blaufox AD, Singh HR, Ross BA, Wong KK, Bar-Cohen Y, McCrindle BW, Etheridge SP. The study of antiarrhythmic medications in infancy (SAMIS): a multicenter, randomized controlled trial comparing the efficacy and safety of digoxin versus propranolol for prophylaxis of supraventricular tachycardia in infants. Circ Arrhythm Electrophysiol. 2012 Oct;5(5):984-91. doi: 10.1161/CIRCEP.112.972620. Epub 2012 Sep 8. PMID 22962431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between December 2006 and August 2010. 14 centers enrolled study participants. Only 72 of the desired 220 subjects enrolled. Enrolment closed early as an independent, unblinded verification of the results determined that a much larger sample size than estimated was necessary to demonstrate the primary outcome existed.
Groups:
- Digoxin: The study drug was given for 6 months or until one of the study end points was reached. To account for differences in pharmacokinetics, the first 2 doses of digoxin were administered oraly at 0.010 mg/kg per dose TID, then 0.0035 mg/kg per dose TID for the third and subsequent doses.
- Propranolol: The study drug was given for 6 months or until one of the study end points was reached. To account for differences in pharmacokinetics, the drug was administered orally at 0.5 mg/kg per dose as a single dose and increased to 1.0 mg/kg per dose TID for the second and subsequent doses.
Period: Overall Study
Arm/Group | Digoxin | Propranolol
Started | 33 | 39
Completed | 27 | 34
Not Completed | 6 | 5
Not completed — Renal impairment | 1 | 0
Not completed — Physician Decision | 5 | 5

BASELINE CHARACTERISTICS:
Population: As 1 subject withdrew after being randomized to digoxin due to renal impairment and did not receive the study drug, the baseline analysis including age continuous data were assessed at enrolment with 32 study participants on digoxin and 39 participants on propranolol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Digoxin | Propranolol | Total
Number analyzed (Participants) | 32 | 39 | 71
Age, Continuous [Median (Full Range); unit: days] | 16.5 [0 to 67] | 7 [0 to 126] | 11.75 [0 to 126]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 23 | 24 | 47
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 34 | 59
  Hispanic/Latino | 2 | 2 | 4
  Black | 3 | 1 | 4
  Native American | 2 | 0 | 2
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Recurrent Supraventricular Tachycardia (SVT) Requiring Medical Intervention to Terminate the Episode.
Time Frame: 6 months or until study endpoints were reached
Measure: Number; unit: percentage of participants
Groups:
- Digoxin: The first 2 doses of digoxin were administered orally at 0.010 mg/kg per dose TID, then 0.0035 mg/kg per dose TID for the third and subsequent doses.
- Propranolol: Single dose administered at 0.5 mg/kg per dose as a single dose and increased to 1.0 mg/kg per dose TID for the second and subsequent doses.
Arm/Group | Digoxin | Propranolol
Number analyzed (Participants) | 32 | 39
percentage of participants | 12 | 18

2. Secondary Outcome: Number of Treated Patients Experiencing First SVT Recurrence
Description: Infants treated with propranolol or digoxin
Time Frame: up to 110 days of treatment
Measure: Number; unit: participants
Groups:
- Propranolol: Single dose administered orally at 0.5/kg per dose and increased to 1.0 mg/kg per dose TID for the second and subsequent doses.
Arm/Group | Digoxin | Propranolol
Number analyzed (Participants) | 32 | 39
participants | 6 | 12 [0.60 to 4.26]

3. Secondary Outcome: Incidence of Adverse Outcomes in Infants With Propranolol or Digoxin
Description: In relation to the study drugs
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Digoxin | Propranolol
Number analyzed (Participants) | 32 | 39
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Digoxin | Propranolol
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/34
Other Adverse Events (participants affected / at risk) | 0/27 | 0/34

LIMITATIONS AND CAVEATS:
Besides issues of recruitment, potential limitations of this study include the selected dosing for propranol, as a higher dosage is sometimes used, and the lack of dose titration before the 2-month visit, both of which could influence drug efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes